CLINICAL TRIAL: NCT06910800
Title: Indwelling Pleural Catheters: Co-developing an Intervention to Support Self-Management
Brief Title: Indwelling Pleural Catheters: a Self-management Intervention
Acronym: PACMAN
Status: Enrolling by invitation | Type: Observational
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Collaborators: University of East Anglia (Other)
Responsible Party: Sponsor
Other Study IDs: Pac-man protocol | v1.0 | 14.0; 333923 (Registry Identifier: IRAS); 58382 (Registry Identifier: CPMS)
Record Dates: First submitted 2025-03-12; First posted 2025-04-04 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Indwelling Pleural Catheter
Keywords: Indwelling pleural catheter; Tunnelled pleural catheter; IPC; Pleural effusion; Self-management; Support needs
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients: Patients who have (or have had) an IPC.
- Family members and unpaid carers: Family members and unpaid carers of patients who have (or have had) an IPC.
- Healthcare professionals: Community nurses involved in IPC care and healthcare professionals involved in IPC insertion.

SUMMARY:
A pleural effusion is a build-up of fluid around the lung. In the UK, about quarter of a million people develop a pleural effusion each year. They are usually caused by advanced cancer or heart, kidney, or liver failure. People with a pleural effusion feel breathless and can't do the things they want to. Draining the fluid improves breathlessness and quality of life. This can be done by inserting a semi-permanent tube called an indwelling pleural catheter (IPC). This is drained at home about three times a week.

Drainage is usually done by a community nurse. However, it can be done by the patient or family/unpaid carers - this is called self-management. Self-management gives the patient the freedom to drain their IPC when they need to, without having to wait at home until a nurse is available. It reduces the burden on community nursing services. Despite these benefits, not all patients get the opportunity to self-manage.

The aim of this study is to help more patients self-manage if they want to. We will achieve this through three stages:

Stage 1: We will talk to patients with IPCs as well as their families/carers to find out their views on self-management and what stops people who could self-manage from doing so. We know that patients with an IPC can be frail. Often their families/carers are already doing a lot to support them. We will ask what might help them to self-manage if they would like to.

Stage 2: We will talk to healthcare professionals (HCPs) looking after patients with IPCs to understand what they think about self-management. This will include community nurses and the hospital teams who put IPCs in.

Stage 3: Along with our patients, their families/unpaid carers and HCPs, we will hold workshops to design an intervention that will help people to self-manage IPCs. We don't know what this intervention will look like yet. From talking to patients and families who already self-manage, we have found they like to learn from a demonstration on their own IPC followed by supervised self-management until they feel confident. Therefore, our intervention may include training sessions for HCPs on how to teach self-management.

This study grew from conversations with our patients. People with an IPC, family members and community nurses helped design the study. Our patient and public involvement (PPI) group will help design study materials and guide the study.

DETAILED DESCRIPTION:
Research question:

How can patients with an indwelling pleural catheter (IPC) and their family/unpaid carers be supported to self-manage?

Background:

Pleural effusion is the accumulation of fluid in the space between the lung and chest wall. It is a common complication of malignancy and affects approximately 200-250,000 people annually in the UK. People with such an effusion experience disabling breathlessness; this is treated by draining the fluid using IPCs (semi-permanent chest drains). These are usually managed at home by community nurses, but this can be done by the patient, family member or carer. Supported self-management is part of the NHS long term plan and British Thoracic Society guidelines state that patients should be supported to self-manage their IPC to promote independence. However, there is no evidence to support these recommendations, nor guidance on how self-management should be facilitated. There is thus an evidence gap at the heart of current recommendations.

Objectives:

O1. Identify support needs of patients with IPCs and their family/unpaid carers and how these impact on the acceptability and feasibility of self-management.

O2. Identify barriers and motivators to IPC self-management among patients and family/unpaid carers.

O3. Understand healthcare professional (HCP) attitudes toward, and practices related to, IPC self-management.

O4. Co-design and develop an evidence-based intervention to facilitate IPC self-management.

Methods:

An applied qualitative study and co-design project comprising three stages mapped to the four objectives.

S1: semi-structured interviews with patients with an IPC and their family/unpaid carers regarding self-management and support needs.

S2: focus groups and interviews with community nurses and IPC service staff regarding self-management.

S3: co-design and development of a self-management intervention.

Interviews will be audio- or audiovisual-recorded (with permission), transcribed, and analysed using thematic analysis. Codes will be assigned to text to categorise meanings. Given the lack of prior research, the coding schema will be developed inductively from early transcripts (with reference to literature from other fields), refined and applied to subsequent transcripts. Codes will be categorised, themes identified, and the results developed into a narrative. The COM-B system will be the model of reference for the development of the self-management intervention. This is comprised of a behaviour change wheel linked to intervention functions and policy categories.

Inclusion criteria Stage 1 - patients and family/unpaid carers

* Adult (>18 years) who has (or has had) an IPC OR
* Adult family member or unpaid carer of a patient who has (or has had) an IPC
* Patients may currently be self-managing or receiving CN care. Stage 2 - healthcare professionals
* Community nurse: experience of caring for a patient with an IPC within the last 12 months and signed-off as competent in IPC management
* IPC-insertion site staff: any HCP involved in discussion with patients about post-insertion IPC care Stage 3 - co-design groups
* as above

Exclusion criteria Stage 1 - patients

* Patient with a life expectancy of less than 6 weeks
* Patient or family/unpaid carer who lacks capacity to offer informed consent (as judged by a suitably qualified HCP in accordance with Good Clinical Practice guidelines) Stage 2 - Health care professionals
* None Stage 3 - co-design groups
* As above

Anticipated Impact and Dissemination

The principal output will be a prototype self-management intervention for patients with an IPC and their family/unpaid carers that will:

* Empower patients, increase perceived symptom control, and reduce time spent 'waiting in' for nursing visits;
* Relieve pressure on community nursing services and reduce healthcare costs;
* Support the NHS long term plan by enabling supported self-management;
* Facilitate more frequent drainage which may prevent re-accumulation of pleural fluid.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1 - Patients and family/unpaid carers

  * Adult (>18 years) who has (or has had) an IPC OR
  * Adult family member or unpaid carer of a patient who has (or has had) an IPC
  * Patients may currently be self-managing or receiving CN care.

Stage 2 - Healthcare professionals

* Community nurse: experience of caring for a patient with an IPC within the last 12 months and signed-off as competent in IPC management
* IPC-insertion site staff: any HCP involved in discussion with patients about post-insertion IPC care

Stage 3 - Co-design groups

o as above

Exclusion Criteria:

* Stage 1 - Patients

  * Patient with a life expectancy of less than 6 weeks
  * Patient or family/unpaid carer who lacks capacity to offer informed consent (as judged by a suitably qualified HCP in accordance with Good Clinical Practice guidelines)

Stage 2 - Health care professionals o None

Stage 3 - Co-design groups

o As above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UK patients who have (or have had) an indwelling pleural catheter, and their family/unpaid carers. UK healthcare professionals who work with patients who have IPCs, including community nurses and IPC-insertion centre staff.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Capturing Health Care Professionals attitudes toward and beliefs about self-management | Periprocedural
  Data will be collected via focus groups and interviews. The different data collection designs reflect the nature of how the two groups of HCPs work and working patterns. The topic guide for the two activities will thus be largely the same and given the common subject matter it will be possible to analyse the qualitative data from these two approaches together. There will be some additional, group-specific, questions reflecting the different roles these two HCP groups play in the patient care pathway.
  The four objectives to achieve this are:
  1. to identify support needs in relation to IPC and how unfulfilled needs impact ability to self-manage.
  2. to identify barriers and motivators to IPC self-management among patients and family/unpaid carers.
  3. to understand HCP attitudes toward, and practices related to, IPC-self-management.
  4. to work with stakeholders to co-develop an intervention to facilitate IPC self-management.

CONTACTS AND LOCATIONS:
Overall Officials: Adam M Dr Peel, Principal Investigator — Norfolk and Norwich University Hospitals NHS Trust
Locations (1):
- Norfolk and Norwich University Hospitals NHS Trust, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The study will be publicised to stakeholders. Online resources may be hosted and promoted via the MyPleuralEffusionJourney and UKPS websites. Further opportunities for promotion will be explored including direct contact with services previously identified as using self-management infrequently.
Supporting Information: CSR
Time Frame: Throughout study duration.
Access Criteria: Stakeholders including - but not limited to:
  * Regional integrated care boards, and participating NHS trusts / study recruitment sites.
  * Influential third sector organisations such as Mesothelioma UK
  * IPC manufacturers
  * Relevant charities such as Breast Cancer UK and the Roy Castle lung cancer foundation.
  * Via the FutureNHS platform.
  * Members of the BTS Pleural Guideline Development group